CLINICAL TRIAL: NCT03239600
Title: A Two Part Phase IIa Study, to Evaluate the Safety and Tolerability, Pharmacokinetics, Proof of Mechanism and Potential for Efficacy of an Anti-IL-7 Receptor-α Monoclonal Antibody (GSK2618960) in the Treatment of Primary Sjögren's Syndrome
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), Proof of Mechanism of GSK2618960 in Primary Sjögren's Syndrome (pSS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is stopped for Portfolio prioritization.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201579
Record Dates: First submitted 2017-06-19; First posted 2017-08-04 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Autoimmune Diseases
Keywords: Anti-IL-7 Receptor-alpha Monoclonal Antibody; Safety; GSK2618960; Primary Sjögren's Syndrome
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2618960; Methotrexate

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment where in Part II of the study, randomized subject will receive GSK2618960 and placebo drug simultaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double blind (sponsor unblind) study and masking will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I & II: GSK2618960 2 milligram per kilogram (mg/kg) (Experimental): GSK2618960 2mg/kg will be administered intravenously (IV) with Methotrexate (MTX)
  Interventions: Drug: GSK2618960 2 mg/kg; Drug: Methotrexate
- Part II: Placebo (Placebo Comparator): Placebo will be administered IV with MTX
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: GSK2618960 2 mg/kg — GSK2618960 solution for injection, 100mg/mL is clear to opalescent, colorless to yellow or pale brown liquid.
  Arms: Part I & II: GSK2618960 2 milligram per kilogram (mg/kg)
Drug: Placebo — Placebo solution will be administered by IV infusion.
  Arms: Part II: Placebo
Drug: Methotrexate — MTX dose between 7.5 to 15 mg will be administered in tablet form once in a week till last dose of GSK2618960 to all subjects in Part I and Part II.

SUMMARY:
This study aims to evaluate the safety, tolerability and PK of repeat dose administration of GSK2618960 in the treatment of pSS. The study will contain two parts, Part I will be open label and Part II will be randomized, double-blind. The minimum duration of Part I & Part II of the study will be 26 and 32 weeks respectively.

ELIGIBILITY:
Inclusion Criteria:

* Part I and Part II: Male and females aged 18-70
* Part I and Part II: pSS diagnosis according to the American-European Consensus Group Criteria
* Part I and Part II: Documented previous biopsy evidence of salivary gland inflammation consistent with pSS and/or documented history of anti-Ro and/or anti-La antibodies
* Part II: Has any of the following abnormalities at screening: hypergammaglobulinaemia [serum Immunoglobulin G (IgG) greater than or equal to 16 gram per liter (g/L); Presence of Rheumatoid factor (RF); Anti Nuclear Antibodies (ANA) titer greater than or equal to 320:1.
* Stimulated whole salivary flow greater than 0.1 milliliter per minute (mL/min) at screening.
* Symptomatic oral dryness greater than or equal to 5 out of 10 on Visual Analogue Scale (VAS) scale and/or Schirmer test less than 10 millimeter (mm) at screening.

Exclusion Criteria:

* Part I and II: Secondary Sjögren's Syndrome
* Part I and II: Receiving cyclophosphamide, other biologic, immunosuppressive or immunomodulatory treatments
* Part I and II: Active infections, or history of recurrent infections
* Part I and II: History of significant medical illness
* Part I and II: History of lymphoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AEs): Part 1 | Up to Week 29
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Number of subjects with abnormal clinical chemistry values: Part 1 | Up to Week 29
  Samples for clinical chemistry tests will be collected as a measure of safety
Number of subjects with abnormal hematology values: Part 1 | Up to Week 29
  Samples for clinical hematology tests will be collected as a measure of safety
Number of subjects with abnormal urine analysis values: Part 1 | Up to Week 29
  Samples for Urine analysis tests will be collected as a measure of safety
Number of subjects with abnormal findings of body temperature: Part 1 | Up to Week 29
  Body temperature will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of blood pressure: Part 1 | Up to Week 29
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of pulse rate: Part 1 | Up to Week 29
  Pulse rate will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of respiratory rate: Part 1 | Up to Week 29
  Respiratory rate will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal Electrocardiogram (ECG) findings: Part 1 | Up to Week 29
  Triplicate 12-lead ECGs will be obtained at each time point using an ECG machine
Number of subjects with AEs: Part 2 | Up to Week 35
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Number of subjects with abnormal clinical chemistry values: Part 2 | Up to Week 35
  Samples for clinical chemistry tests will be collected as a measure of safety
Number of subjects with abnormal hematology values: Part 2 | Up to Week 35
  Samples for clinical hematology tests will be collected as a measure of safety
Number of subjects with abnormal urine analysis values: Part 2 | Up to Week 35
  Samples for Urine analysis tests will be collected as a measure of safety
Number of subjects with abnormal findings of body temperature: Part 2 | Up to Week 35
  Body temperature will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of blood pressure: Part 2 | Up to Week 35
  SBP and DBP will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of pulse rate: Part 2 | Up to Week 35
  Pulse rate will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal findings of respiratory rate: Part 2 | Up to Week 35
  Respiratory rate will be measured in a semi-supine position after at least a 5-minute rest.
Number of subjects with abnormal ECG findings: Part 2 | Up to Week 35
  Triplicate 12-lead ECGs will be obtained at each time point using an ECG machine

SECONDARY OUTCOMES:
Plasma concentration of GSK2618960: Part 1 | Day 1: post-infusion; Day 15 and 29: pre-infusion; Day 43: Pre and post-infusion; Day 8, 22, 36, 50, 57, 71, 99 and 127
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters.
Maximum observed plasma concentration (Cmax) of GSK2618960: Part 1 | Day 1: post-infusion; Day 15 and 29: pre-infusion; Day 43: Pre and post-infusion; Day 8, 22, 36, 50, 57, 71, 99 and 127
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters.
Minimum observed plasma concentration (Cmin) of GSK2618960: Part 1 | Day 1: post-infusion; Day 15 and 29: pre-infusion; Day 43: Pre and post-infusion; Day 8, 22, 36, 50, 57, 71, 99 and 127
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters.
Area under the curve (AUC) of GSK2618960: Part 1 | Day 1: post-infusion; Day 15 and 29: pre-infusion; Day 43: Pre and post-infusion; Day 8, 22, 36, 50, 57, 71, 99 and 127
  Blood samples will be collected prior to start and at the end of infusion at indicated time points and will be analyzed for PK parameters.
Number of incidences of Anti-drug antibody (ADA) formation: Part 1 | Up to Week 29
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Number of titres of ADA: Part 1 | Up to Week 29
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Time to onset of ADA: Part 1 | Up to Week 29
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Number of incidences of ADA neutralization: Part 1 | Up to Week 29
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Plasma concentration of GSK2618960 : Part 2 | Day 1: post-infusion; Day 15, 29, 43, 57: pre-infusion; Day 71: Pre and post-infusion; Day 8, 22, 36, 50, 64, 78, 85, 113 and 169
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters
Cmax of GSK2618960: Part 2 | Day 1: post-infusion; Day 15, 29, 43, 57: pre-infusion; Day 71: Pre and post-infusion; Day 8, 22, 36, 50, 64, 78, 85, 113 and 169
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters.
Cmin of GSK2618960: Part 2 | Day 1: post-infusion; Day 15, 29, 43, 57: pre-infusion; Day 71: Pre and post-infusion; Day 8, 22, 36, 50, 64, 78, 85, 113 and 169
  Blood samples will be collected prior to start and at the end of infusion at the indicated time points and will be analyzed for PK parameters.
AUC of GSK2618960: Part 2 | Day 1: post-infusion; Day 15, 29, 43, 57: pre-infusion; Day 71: Pre and post-infusion; Day 8, 22, 36, 50, 64, 78, 85, 113 and 169
  Blood samples will be collected prior to start and at the end of infusion at indicated time points and will be analyzed for PK parameters.
Number of incidences of ADA formation: Part 2 | Up to Week 35
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Number of titres of ADA: Part 2 | Up to Week 35
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Time to onset of ADA: Part 2 | Up to Week 35
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Number of incidences of ADA neutralization: Part 2 | Up to Week 35
  Serum samples will be collected from subjects prior to infusion and various time points post-infusion to carry out immunogenicity and immune-complex analyses.
Receptor occupancy (RO) on circulating T cells: Part 2 | Up to Week 35
  Blood samples will be collected from subjects at indicated time points to measure IL-7R alpha occupancy levels.
Percentage inhibition of Signal transducer and activator of transcription 5 (STAT 5) phosphorylation in T cells: Part 2 | Up to Week 35
  Blood samples will be collected from subjects at indicated time points to measure phosphorylation of STAT 5 in response to ex vivo IL-7 stimulation.
Change from Baseline in Focus score: Part 2 | Up to Day 29
  Salivary glands for immunohistochemistry analysis will be evaluated for general appearance and total inflammatory infiltrate (focus score). Salivary gland biopsy will be performed at Baseline and blood samples will be collected at indicated time points.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom